CLINICAL TRIAL: NCT00240383
Title: A Randomized, Double-Blind, Dose Ranging, Dose Comparison-Controlled Trial to Determine the Safety and Efficacy of BMS-298585 in Subjects With Type 2 Diabetes
Brief Title: Dose Ranging Study With LT, Monotherapy, PPAR
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV168-006
Record Dates: First submitted 2005-10-17; First posted 2005-10-18 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2008-06

CONDITIONS: Diabetes Mellitus II
MeSH Terms: interventions — muraglitazar

INTERVENTIONS:
Drug: Muraglitazar

SUMMARY:
A Randomized, Double-Blind, Dose-Ranging, Dose Comparison-Controlled Trial to Determine the Safety and Efficacy of BMS-298585 in Subjects with Type 2 Diabetes

ELIGIBILITY:
Inclusion Criteria:

* 1. HbA1c > 7.0% and ≤ 10.0% obtained at the Screening visit.
* 2. Men and women, 18-70 years of age Established Type 2 diabetes

Exclusion Criteria:

* 1. Symptomatic Type 2 diabetes defined as marked polyuria and polydipsia with greater than 10% weight loss during the last three months.
* 2. Administration of antihyperglycemic agents (other than thiazolidinediones) for more than three consecutive or a total of seven non-consecutive days during the four weeks prior to screening.
* 3. Administration of thiazolidinediones for more than three consecutive or a total of seven non-consecutive days during the six weeks prior to screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1260
Dates: Start 2002-05; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
To compare, after 24 weeks of oral administration of double-blind treatment, the change from baseline in hemoglobin A1c (HbA1c) achieved with the highest dose and subsequent doses of BMS-298585 versus the lowest dose of BMS-298585 in subjects with Type 2

SECONDARY OUTCOMES:
To assess, after 12 and 24 weeks of oral administration of double-blind therapy, the percent change from baseline in fasting lipids (total cholesterol,low density lipoprotein cholesterol,HDL-C, TG, non-HDL chol

CONTACTS AND LOCATIONS:
Locations (272):
- United States (149):
  - Local Institution, Anniston, Alabama
  - Local Institution, Birmingham, Alabama
  - Local Institution, Huntsville, Alabama
  - Local Institution, Hot Springs, Arizona
  - Local Institution, Mesa, Arizona
  - Local Institution, Phoenix, Arizona
  - Local Institution, Tempe, Arizona
  - Local Institution, Tucson, Arizona
  - Local Institution, Fayette, Arkansas
  - Local Institution, Little Rock, Arkansas
  - Local Institution, Bakersfield, California
  - Local Institution, Concord, California
  - Local Institution, Encinitas, California
  - Local Institution, Fair Oaks, California
  - Local Institution, Fountain Valley, California
  - Local Institution, Fresno, California
  - Local Institution, La Jolla, California
  - Local Institution, Los Gatos, California
  - Local Institution, Orange, California
  - Local Institution, Raleigh, California
  - Local Institution, Riverside, California
  - Local Institution, Rolling Hills Estate, California
  - Local Institution, Roseville, California
  - Local Institution, Sacramento, California
  - Local Institution, San Diego, California
  - Local Institution, Santa Ana, California
  - Local Institution, Santa Barbara, California
  - Local Institution, Spring Valley, California
  - Local Institution, Tustin, California
  - Local Institution, Walnut Creek, California
  - Local Institution, Colorado Springs, Colorado
  - Local Institution, Golden, Colorado
  - Local Institution, Littleton, Colorado
  - Local Institution, Nederland, Colorado
  - Local Institution, Wheat Ridge, Colorado
  - Local Institution, New Britain, Connecticut
  - Local Institution, Brandon, Florida
  - Local Institution, Chipley, Florida
  - Local Institution, Coral Gables, Florida
  - Local Institution, Daytona Beach, Florida
  - Local Institution, Fort Lauderdale, Florida
  - Local Institution, Hollywood, Florida
  - Local Institution, Jacksonville, Florida
  - Local Institution, Jupiter, Florida
  - Local Institution, Melbourne, Florida
  - Local Institution, Miami, Florida
  - Local Institution, Ocala, Florida
  - Local Institution, Ocoee, Florida
  - Local Institution, Orlando, Florida
  - Local Institution, Pensacola, Florida
  - Local Institution, St. Petersburg, Florida
  - Local Institution, Tallahassee, Florida
  - Local Institution, Tamarac, Florida
  - Local Institution, Titusville, Florida
  - Local Institution, West Palm Beach, Florida
  - Local Institution, Atlanta, Georgia
  - Local Institution, Dunwoody, Georgia
  - Local Institution, Honolulu, Hawaii
  - Local Institution, Chicago, Illinois
  - Local Institution, Vernon Hills, Illinois
  - Local Institution, Arkansas City, Kansas
  - Local Institution, Shawnee Mission, Kansas
  - Local Institution, Wichita, Kansas
  - Local Institution, Bardstown, Kentucky
  - Local Institution, Lexington, Kentucky
  - Local Institution, Louisville, Kentucky
  - Local Institution, Richmond, Kentucky
  - Local Institution, Metairie, Louisiana
  - Local Institution, Slidell, Louisiana
  - Local Institution, Bangor, Maine
  - Local Institution, Baltimore, Maryland
  - Local Institution, Chevy Chase, Maryland
  - Local Institution, Norwood, Massachusetts
  - Local Institution, Springfield, Massachusetts
  - Local Institution, Swansea, Massachusetts
  - Local Institution, Worcester, Massachusetts
  - Local Institution, Birmingham, Michigan
  - Local Institution, Petoskey, Michigan
  - Local Institution, Arden Hills, Minnesota
  - Local Institution, Bay Saint Louis, Mississippi
  - Local Institution, Cleveland, Mississippi
  - Local Institution, Jackson, Mississippi
  - Local Institution, Olive Branch, Mississippi
  - Local Institution, Rolling Fork, Mississippi
  - Local Institution, Excelsior Springs, Missouri
  - Local Institution, Kansas City, Missouri
  - Local Institution, Springfield, Missouri
  - Local Institution, St Louis, Missouri
  - Local Institution, Omaha, Nebraska
  - Local Institution, Las Vegas, Nevada
  - Local Institution, Toms River, New Jersey
  - Local Institution, Albuquerque, New Mexico
  - Local Institution, Buffalo, New York
  - Local Institution, Camillus, New York
  - Local Institution, Endicott, New York
  - Local Institution, Johnson City, New York
  - Local Institution, New Hyde Park, New York
  - Local Institution, New York, New York
  - Local Institution, Cary, North Carolina
  - Local Institution, Charlotte, North Carolina
  - Local Institution, Greensboro, North Carolina
  - Local Institution, High Point, North Carolina
  - Local Institution, Moorehead City, North Carolina
  - Local Institution, Raleigh, North Carolina
  - Local Institution, Avon, Ohio
  - Local Institution, Beavercreek, Ohio
  - Local Institution, Bellbrook, Ohio
  - Local Institution, Canton, Ohio
  - Local Institution, Cincinnati, Ohio
  - Local Institution, Cleveland, Ohio
  - Local Institution, Colombus, Ohio
  - Local Institution, Lyndhurst, Ohio
  - Local Institution, Massillon, Ohio
  - Local Institution, Zanesville, Ohio
  - Local Institution, Tulsa, Oklahoma
  - Local Institution, Eugene, Oregon
  - Local Institution, Medford, Oregon
  - Local Institution, Portland, Oregon
  - Local Institution, Reading, Pennsylvania
  - Local Institution, Cranston, Rhode Island
  - Local Institution, East Providence, Rhode Island
  - Local Institution, Johnston, Rhode Island
  - Local Institution, Providence, Rhode Island
  - Local Institution, Anderson, South Carolina
  - Local Institution, Charleston, South Carolina
  - Local Institution, Greer, South Carolina
  - Local Institution, Simpsonville, South Carolina
  - Local Institution, Spartanburg, South Carolina
  - Local Institution, Bristol, Tennessee
  - Local Institution, Johnson City, Tennessee
  - Local Institution, Memphis, Tennessee
  - Local Institution, Austin, Texas
  - Local Institution, Corpus Christi, Texas
  - Local Institution, Dallas, Texas
  - Local Institution, Fort Worth, Texas
  - Local Institution, Houston, Texas
  - Local Institution, Irving, Texas
  - Local Institution, Lake Jackson, Texas
  - Local Institution, San Antonio, Texas
  - Local Institution, Salt Lake City, Utah
  - Local Institution, Richmond, Virginia
  - Local Institution, Virginia Beach, Virginia
  - Local Institution, Edmonds, Washington
  - Local Institution, Federal Way, Washington
  - Local Institution, Renton, Washington
  - Local Institution, Spokane, Washington
  - Local Institution, Walla Walla, Washington
  - Local Institution, Madison, Wisconsin
  - Local Institution, New Berlin, Wisconsin
- Argentina (3):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Chacabuco, Buenos Aires
  - Local Institution, Mendoza, Mendoza Province
- Australia (7):
  - Local Institution, Wollongong, New South Wales
  - Local Institution, Fullerton, South Australia
  - Local Institution, Box Hill, Victoria
  - Local Institution, Fitzroy, Victoria
  - Local Institution, Melbourne, Victoria
  - Local Institution, Parkville, Victoria
  - Local Institution, Perth, Western Australia
- Brazil (10):
  - Local Institution, Fortaleza, Ceará
  - Local Institution, Campo Grande, Mato Grosso
  - Local Institution, Belém, Pará
  - Local Institution, Rio de Janeiro, Rio de Janeiro
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Campinas, São Paulo
  - Local Institution, Marília, São Paulo
  - Local Institution, S. J. Rio Preto, São Paulo
  - Local Institution, São Paulo, São Paulo
  - Local Institution, Taubaté, São Paulo
- Canada (9):
  - Local Institution, Calgary, Alberta
  - Local Institution, Edmonton, Alberta
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, St. John's, Newfoundland and Labrador
  - Local Institution, Ottawa, Ontario
  - Local Institution, Drummonville, Quebec
  - Local Institution, Longueuil, Quebec
  - Local Institution, Ottawa, Quebec
  - Local Institution, Sherbrooke, Quebec
- Czechia (5):
  - Local Institution, Brno, CZE
  - Local Institution, České Budějovice
  - Local Institution, Jihlava
  - Local Institution, Liberec
  - Local Institution, Prague
- France (6):
  - Local Institution, Albens
  - Local Institution, Orthez
  - Local Institution, Rennes
  - Local Institution, Rosiers-d'Égletons
  - Local Institution, Savigny-en-Véron
  - Local Institution, Strasbourg
- Italy (3):
  - Local Institution, Milan
  - Local Institution, Modena
  - Local Institution, Roma
- Mexico (4):
  - Local Institution, Aguascalientes, Aguascalientes
  - Local Institution, Tijuana, Estado de Baja California
  - Local Institution, Distrito Federal, Mexico City
  - Local Institution, Mexico City, Mexico City
- Netherlands (7):
  - Local Institution, Deventer
  - Local Institution, Ewijk
  - Local Institution, Hengelo
  - Local Institution, Lichtenvoorde
  - Local Institution, Losser
  - Local Institution, Ryswyk
  - Local Institution, Utrecht
- Poland (10):
  - Local Institution, Gorzów, Wielkopolski
  - Local Institution, Stalowa, Wola
  - Local Institution, Bydgoszcz
  - Local Institution, Lublin
  - Local Institution, Olsztyn
  - Local Institution, Szczecin
  - Local Institution, Warsaw
  - Local Institution, Wroclaw
  - Local Institution, Zabrze
  - Local Institution, Zielona Góra
- Puerto Rico (2):
  - Local Institution, Ponce
  - Local Institution, San Juan
- South Africa (5):
  - Local Institution, Noordheuwel, Gauteng
  - Local Institution, Pretoria, Gauteng
  - Local Institution, Vanderbijlpark, Gauteng
  - Local Institution, George, Northern Cape
  - Local Institution, Tygerberg, Western Cape
- Spain (9):
  - Local Institution, Santiago, De Compostela
  - Local Institution, Barcelona, ESP
  - Local Institution, Cadiz, ESP
  - Local Institution, Herston, Queensland
  - Local Institution, Girona
  - Local Institution, Granada
  - Local Institution, Las Palmas de Gran Canaria
  - Local Institution, Madrid
  - Local Institution, Oviedo
- Sweden (8):
  - Local Institution, Gothenburg
  - Local Institution, Helsingborg
  - Local Institution, Linköping
  - Local Institution, Malmo
  - Local Institution, Motala
  - Local Institution, Sävedalen
  - Local Institution, Stockholm
  - Local Institution, Vällingby
- United Kingdom (35):
  - Local Institution, Newtonabbey, Armach
  - Local Institution, Ely, Cambridgeshire
  - Local Institution, Soham, Cambridgeshire
  - Local Institution, Blantyre, Central
  - Local Institution, Chapelhall, Central
  - Local Institution, Paisley, Central
  - Local Institution, Riddrie, Central
  - Local Institution, Cumbernauld, Dumbartonshire
  - Local Institution, Moodiesburn, Dumbartonshire
  - Local Institution, Annan, Dumfries & Galloway
  - Local Institution, Dunscore, Dumfries & Galloway
  - Local Institution, Stranraer, Dumfries & Galloway
  - Local Institution, Moffat, Dumfriesshire
  - Local Institution, Bexhill-on-Sea, East Sussex
  - Local Institution, High Valleyfield, Fife
  - Local Institution, Sunbury-on-Thames, Greater London
  - Local Institution, Caerleon, Gwent
  - Local Institution, Burnbank, Lanarkshire
  - Local Institution, Coatbridge, Lanarkshire
  - Local Institution, Edinburgh, Lothian
  - Local Institution, Hamilton, Lothian
  - Local Institution, Llandough, Mid Glamorgan
  - Local Institution, Pont-y-clun, Mid Glamorgan
  - Local Institution, Neilston, Renfrewshire
  - Local Institution, Paisley, Renfrewshire
  - Local Institution, Kilsyth, Stirlingshire
  - Local Institution, Lanarkshire, Strathclyde
  - Local Institution, East Horsley, Surrey
  - Local Institution, Cookstown, Tyrone
  - Local Institution, Atherstone, Warwickshire
  - Local Institution, Balsall Common, Warwickshire
  - Local Institution, Stratford-upon-Avon, Warwickshire
  - Local Institution, Chelmsley Wod, West Midlands
  - Local Institution, Chippenham, Wiltshire
  - Local Institution, Glasgow

REFERENCES:
- [Derived] Rubin CJ, Viraswami-Appanna K, Fiedorek FT. Efficacy and safety of muraglitazar: a double-blind, 24-week, dose-ranging study in patients with type 2 diabetes. Diab Vasc Dis Res. 2009 Jul;6(3):205-15. doi: 10.1177/1479164109336048. PMID 20368213